CLINICAL TRIAL: NCT07383142
Title: Surgery Combined With Hyperthermic Intrathoracic Chemotherapy Versus Surgery Alone for Pleural Dissemination or Pleural Recurrence of Thymic Epithelial Tumors: A Prospective, Multicenter, Randomized Controlled Clinical Trial
Brief Title: Intrathoracic Chemotherapy for TETs With Pleural Spread or Recurrence (CHOICE-2)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Sir Run Run Shaw Hospital (Other); West China Hospital (Other); Liaoning Cancer Hospital & Institute (Other); Fujian Medical University Union Hospital (Other); Qilu Hospital of Shandong University (Other); Jiangxi Provincial People's Hopital (Other); Zhongshan Hospital (Xiamen), Fudan University (Other); Tang-Du Hospital (Other); Xuhui Central Hospital, Shanghai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHOICE-2
Record Dates: First submitted 2026-01-14; First posted 2026-02-03 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Thymic Epithelial Tumor
Keywords: Hyperthermic Intrathoracic Chemotherapy
MeSH Terms: conditions — Thymic epithelial tumor | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery alone (Active Comparator)
  Interventions: Procedure: Surgery alone
- Surgery+HITOC (Experimental)
  Interventions: Procedure: Surgery+HITOC

INTERVENTIONS:
Procedure: Surgery alone — Patients undergo lung-preserving cytoreductive surgery, including pleurectomy/decortication (P/D) or extended pleurectomy/decortication (eP/D), via video-assisted thoracoscopic surgery (VATS) or thoracotomy. The goal is to achieve macroscopic complete resection of all visible pleural nodules and involved structures (e.g., pericardium, diaphragm). Extrapleural pneumonectomy (EPP) is excluded from the surgical strategy.
  Arms: Surgery alone
Procedure: Surgery+HITOC — Patients undergo the same cytoreductive surgery (P/D or eP/D) as the control group. Following surgery, patients receive hyperthermic intrathoracic chemotherapy (HITOC) using a hyperthermic perfusion system heated to 43°C. The regimen consists of intrathoracic perfusion with doxorubicin (25 mg/m²) on postoperative day 1 (POD 1), followed by intrathoracic perfusion with cisplatin (50 mg/m²) on postoperative day 2 (POD 2).
  Arms: Surgery+HITOC

SUMMARY:
Hyperthermic intrathoracic chemotherapy (HITOC) offers a strategy to eliminate microscopic residual disease after surgical resection. Especially it is investigated to improve long-term survival in thymic epithelial tumors with pleural dissemination or recurrence. A prospective, multicenter, randomized phase III clinical trial (CHOICE-2) is conducted to compare the efficacy and safety of surgery combined with HITOC versus surgery alone. The HITOC regimen involves intrathoracic perfusion with doxorubicin on postoperative day 1 and cisplatin on postoperative day 2.

DETAILED DESCRIPTION:
Thymic epithelial tumors (TETs) frequently manifest with or recur as pleural dissemination (Stage IVa), presenting a significant clinical challenge. Although cytoreductive surgery is the cornerstone of treatment, achieving complete elimination of microscopic residual disease remains difficult, often leading to subsequent recurrence. Hyperthermic intrathoracic chemotherapy (HITOC) has emerged as a promising adjuvant strategy to control local disease by combining the cytotoxic effects of chemotherapy with hyperthermia to eradicate microscopic residuals.

Building on the favorable safety and efficacy results from the Phase II CHOICE study, the CHOICE-2 study is a prospective, multicenter, randomized, phase III clinical trial designed to compare surgery combined with HITOC versus surgery alone. A total of 202 eligible participants with pleural dissemination or pleural recurrence of TETs will be randomized in a 1:1 ratio into two arms.

Participants in the experimental arm will undergo lung-preserving cytoreductive surgery (pleurectomy/decortication or extended pleurectomy/decortication) followed by HITOC. The HITOC regimen involves intrathoracic perfusion with doxorubicin (25 mg/m²) on postoperative day 1 and cisplatin (50 mg/m²) on postoperative day 2, utilizing a perfusion system heated to 43°C for 60 minutes. Participants in the control arm will receive the same standard surgical resection without HITOC.

The primary objective is to evaluate the 3-year progression-free survival (PFS) rate. Secondary endpoints include overall survival (OS), myasthenia gravis (MG) remission rates according to MGFA criteria, and the incidence of perioperative complications.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18-75 years old; Expected survival time > 12 months; Preoperative imaging (CT, MRI, or PET-CT) clinically diagnosed as TETs
2. Patients with de novo stage IVa thymoma (DNT) diagnosed by the multidisciplinary team (MDT) are eligible if deemed suitable for surgery under any of the following conditions: (1) candidates for primary surgery without contraindications; (2) candidates for staged surgery who have completed phase I surgery and are reassessed by the MDT as eligible for phase II surgery 3 months postoperatively; or (3) patients initially requiring induction therapy, provided the diagnosis is pathologically confirmed by biopsy, induction therapy is administered according to TET guidelines, imaging and laboratory evaluations are performed 4-6 weeks after completion of therapy, and the MDT confirms the absence of surgical contraindications upon re-evaluation.
3. For patients with thymoma with pleural recurrence (TPR), the initial surgery must have achieved complete resection without evidence of pleural dissemination or intraoperative tumor rupture, and the interval between the first surgery and the development of pleural metastasis must be longer than 6 months.
4. According to the definition of T1-3NxM1a stage, no intrapericardial dissemination, no intrapulmonary parenchymal metastatic nodules, no distant organ metastasis (M1b)
5. During the operation, the pleural nodules were removed. The frozen section pathology during the operation confirmed that the pleural nodules were TETs pleural metastatic nodules.
6. No history of other malignant tumors, except for patients who had prior malignancies treated with curative surgery, were confirmed to have pathologic stage I disease requiring no adjuvant therapy (e.g., resected pulmonary ground-glass opacity or papillary thyroid carcinoma) and have remained free of recurrence for more than 5 years.
7. ASA stage I/II
8. Be able to understand the situation of this study and sign the Informed Consent form.

Exclusion Criteria:

1. Preoperative imaging examinations such as CT, MRI or PET-CT, or intraoperative exploration revealed that the tumor involved the ascending aorta, aortic arch, descending aorta, intrapericardial pulmonary vessels, heart, trachea or esophagus (T4), or had dissemination within the pericardium (M1a) or hematogenous metastasis (M1b stage);
2. Within 4-6 weeks after completion of induction therapy (chemotherapy, radiotherapy, immunotherapy, or targeted therapy), imaging studies (CT or PET-CT) and laboratory evaluations (complete blood count, liver and renal function, cardiac biomarkers, and thyroid function) were performed by the mediastinal MDT to assess surgical eligibility; patient found to have surgical contraindications and deemed unsuitable for surgery or HITOC were excluded;
3. The diagnosis was confirmed by biopsy or puncture as a non-TETs type (such as lymphoma, neurogenic tumor, germ cell tumor, thymic lipoma, thymic sarcoma or neuroendocrine tumor);
4. The patient had a history of multiple surgeries in the past (≥2), the initial surgery of TPR was palliative resection, and pleural dissemination was a iatrogenic implantation site; or the patient received a radiotherapy dose greater than 60 Gy before enrollment;
5. Had other active malignant tumors, or had received anti-tumor treatment (chemotherapy, radiotherapy, immunotherapy, small molecule targeted therapy or other anti-tumor biological agents) for other malignant tumors in the past;
6. The patient had myasthenia gravis in an unstable state or during an acute exacerbation;
7. Had the following major cardiovascular disease histories: congestive heart failure, poorly controlled angina pectoris, transmural myocardial infarction, high-risk arrhythmia, significant valvular disease or poorly controlled hypertension, cardiovascular compensatory dysfunction;
8. The patient had a weight loss of more than 5 kg within the past one month; severe uncontrolled systemic systemic diseases, such as active infection or poorly controlled diabetes; patients with bleeding disorders and those with bleeding tendencies; patients with abnormal coagulation function, with bleeding tendencies or undergoing thrombolysis or anticoagulation treatment; patients with grade II-IV bone marrow suppression;
9. The patient had a history of thoracic surgery due to tuberculous pleurisy or mesothelioma, and the contralateral lung atrophy involved one or more lung lobes or more than one lung lobe;
10. The patient had an allergy history to cisplatin or doxorubicin drugs;
11. Had a history of organ transplantation (including autologous bone marrow transplantation and peripheral stem cell transplantation); Had a history of mental disorders, neurological diseases or other central nervous system diseases affecting compliance;
12. The patient was in the acute inflammatory stage due to bacterial, viral or other pathogenic microorganism infection; Had active infection of immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) or known HIV seropositivity;
13. Pregnant or lactating women, and fertile men and women who were unwilling to use adequate contraceptive measures during treatment;
14. The patient had received grade IV surgical treatment within 2 months or was in a recovery state due to other diseases or was in the intervention period of other research projects.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-02-01 (Estimated); Study Completion 2032-02-01 (Estimated)

PRIMARY OUTCOMES:
3-year progression-free survival (PFS) | The 3-year PFS is defined as the proportion of patients who are alive and have not experienced disease progression at 3 years after surgery.

SECONDARY OUTCOMES:
3-year overall survival (OS) | The 3-year OS is defined as the proportion of patients who are alive at 3 years after surgery, regardless of disease status or cause of death.
Myasthenia gravis remission rate (MGFA criteria) | The MG remission rate is calculated at the last follow-up in the three years after surgery.
  The proportion of participants with myasthenia gravis (MG) achieving "Overall Remission" assessed according to the Myasthenia Gravis Foundation of America (MGFA) Post-Intervention Status Classification. As per the study protocol, overall remission is defined as the sum of patients achieving complete stable remission (CSR), pharmacologic remission (PR), or minimal manifestation status (MMS).
Grade ≥3 complications (Clavien-Dindo, 5th ed.) | 1 month postoperatively
  The complication rate was calculated at 1 month after surgery
Quality of life (EORTC QLQ-C30) at 1 month | 1 month postoperatively
Quality of life (EORTC QLQ-C30) at 3 months | 3 months postoperatively
Quality of life (EORTC QLQ-C30) at 6 months | 6 months postoperatively
Perioperative myasthenic crisis incidence | 1 month postoperatively
  Postoperative Myasthenic Crisis (POMC) is defined as respiratory failure caused by myasthenia gravis (MG) requiring immediate intubation and total postoperative ventilatory support for more than 24 hours or requiring re-intubation and ventilatory support within 30 days after extubation. The POMC rate was calculated at 1 month after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No